CLINICAL TRIAL: NCT03154567
Title: Effects of Stress and Drug-cue Exposure on Craving and Marijuana Seeking Behavior in Regular Cannabis Smokers
Brief Title: Effects of Stress and Drug-cue Exposure (SCM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wayne State University (Other)
Responsible Party: Principal Investigator, Leslie Lundahl, Principal Investigator, Wayne State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: SCM-1
Record Dates: First submitted 2017-04-25; First posted 2017-05-16 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Marijuana Abuse
MeSH Terms: conditions — Marijuana Abuse | interventions — Yohimbine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (6):
- Yohimbine 0mg X Cue Condition (neutral) (Placebo Comparator)
  Interventions: Drug: Yohimbine
- Yohimbine 0mg X Cue Condition (marijuana) (Placebo Comparator)
  Interventions: Drug: Yohimbine
- Yohimbine 20mg X Cue Condition (neutral) (Active Comparator)
  Interventions: Drug: Yohimbine
- Yohimbine 20mg X Cue Condition (marijuana) (Active Comparator)
  Interventions: Drug: Yohimbine
- Yohimbine 40mg X Cue Condition (neutral) (Active Comparator)
  Interventions: Drug: Yohimbine
- Yohimbine 40mg X Cue Condition (marijuana) (Active Comparator)
  Interventions: Drug: Yohimbine

INTERVENTIONS:
Drug: Yohimbine — Yohimbine (0mg, 20mg, or 40 mg) will be administered at 11:00am on each of the experimental sessions.

SUMMARY:
The purpose of the proposed study to examine the links among stress, craving for marijuana, and marijuana reminders, or "cues".

In this study, an agent called yohimbine will be used to produce stress-like responses. Yohimbine is known to cause stress response in studies of alcohol and other substance use disorders. This study intends to show it can be used to cause stress in marijuana users as well.

DETAILED DESCRIPTION:
Part of this study will be conducted on a residential unit where participants will live for 7 nights over a 2-week period (4 consecutive nights the 1st week and 3 consecutive nights the 2nd week).

During that time, participants can't leave the unit unescorted or have visitors.

During the inpatient stay participants will participant in experimental sessions where they will be asked to smoke cigarettes containing either marijuana or placebo (a blank).

Participants will be asked to take capsules that could contain yohimbine or placebo (blank).

Participants will be asked to complete questionnaires and will have their vital signs (blood pressure, heart rate) monitored throughout each session.

Participants will be asked to participate in overnight sleep recordings, a polysomnogram (PSG).

ELIGIBILITY:
Inclusion Criteria:

* Participants (18-55 yr) will be current marijuana users, based on self-report and THC-positive urine samples.
* Candidates must meet DSM-5 criteria for Mild-to-Moderate Cannabis Use Disorder (CUD) and be willing to participate in research but not seeking treatment.
* Candidates must be in good health, as assessed using data from psychiatric evaluation, extensive substance use history interview, and medical evaluations including medical history, physical exam, standard lab tests and 12-lead ECG.

Exclusion Criteria:

Candidates with the following conditions will be excluded:

* Serious psychiatric illness (e.g. psychotic or bipolar disorder, recent suicide attempts, major depression).
* Substance Use Disorders other than Cannabis or Nicotine Use Disorders and Mild Alcohol Use Disorder.
* Neurological diseases
* Cardiovascular problems (e.g. including systolic BP >140 or <95 mmHg, diastolic BP >90 mmHg, abnormal ECG).
* Pulmonary diseases
* Systemic diseases
* Cognitive impairment (<80 IQ)
* Past-month medications that increase study risk.
* Women who are pregnant, lactating, or if heterosexually active and not using medically approved birth control.
* Candidates seeking Substance Use Disorder treatment.
* Individuals unable to give voluntary informed consent will be excluded.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2023-10-27 (Actual); Study Completion 2023-10-27 (Actual)

PRIMARY OUTCOMES:
Marijuana Craving Visual Analog Scale (VAS) (Self-report measure) | Change is being assessed. Marijuana Craving VAS administered at baseline 0900. It will then be administered at 1000, 1030, 1100, 1200, 1220, 1245, 1300, 1315, 1345.
Marijuana Craving Questionnaire (Self-report measure) | Change is being assessed. Marijuana Craving Quest.administered at baseline 0900. It will then be administered at 1000, 1030, 1100, 1200, 1410, 1430, 1500, 1530, 1600, 1630.
Questionnaire of Smoking Urges (Self-report measure) | Change is being assessed. Questionnaire is administered at baseline 0900. It will then be administered at 1000, 1030, 1100, 1200, 1410, 1430, 1500, 1530, 1600, 1630.
Marijuana Rating Form (Self-report measure) | Change is being assessed. Marijuana Rating Form is administered 30 minutes after each smoking episode in the sampling session.
Marijuana Withdrawal Checklist | Change is being assessed. Questionnaire is administered every morning and evening.
Subjective Effects Scale Visual Analog Scale (VAS) (Self-report measure) | Change is being assessed. Subjective Effects Scale administered at baseline 0900.It will then be administered at 1000, 1030, 1100, 1200, 1410, 1430, 1500, 1530, 1600, 1630.
Positive & Negative Affect Schedule (Self-report measure) | Change is being assessed. Questionnaire is administered at baseline 0900. It will then be administered at 1000, 1030, 1100, 1200, 1410, 1430, 1500, 1530, 1600, 1630.
Systolic blood pressure (physiological effects) | Change is being assessed. Systolic blood pressure measured at baseline 0900. It will then be measure at 1000, 1030, 1100, 1200, 1410, 1430, 1500, 1530, 1600, 1630.
Diastolic blood pressure (physiological effects) | Change is being assessed. Diastolic blood pressure measured at baseline 0900. It will then be measure at 1000, 1030, 1100, 1200, 1410, 1430, 1500, 1530, 1600, 1630.
Heart rate (physiological effects) | Change is being assessed. Heart rate measured at baseline 0900. It will then be measure at 1000, 1030, 1100, 1200, 1410, 1430, 1500, 1530, 1600, 1630.
Core-body temperature (physiological effects) | Change is being assessed. Core-body temperature measured at baseline 0900. It will then be measure at 1000, 1030, 1100, 1200, 1410, 1430, 1500, 1530, 1600, 1630.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Lundahl, PhD, Principal Investigator — Wayne State University
Locations (1):
- Tolan Park Medical Building, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No